CLINICAL TRIAL: NCT05933109
Title: Augmentation of Imagery Rehearsal Therapy With Targeted Memory Reactivation for Post-Traumatic Stress Disorder (PTSD)
Brief Title: Mental Imagery and Targeted Memory Reactivation in PTSD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Lampros Perogamvros, Attending Physician, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-02270_TR
Record Dates: First submitted 2023-06-20; First posted 2023-07-06 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Nightmares, REM-Sleep Type; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TMR group (Experimental): Patients will receive a sound S1 while they generate a positive outcome of imagery rehearsal therapy (IRT). They will also receive the sound S1 during REM sleep.
  Interventions: Behavioral: Imagery Rehearsal Therapy and Targeted memory reactivation during REM sleep
- Control group (Active Comparator): Patients will not receive the sound S1 while they generate a positive outcome of imagery rehearsal therapy (IRT). During REM sleep, they will receive the same sound as the experimental group (S1) under the same conditions.
  Interventions: Behavioral: Imagery Rehearsal Therapy

INTERVENTIONS:
Behavioral: Imagery Rehearsal Therapy and Targeted memory reactivation during REM sleep — Emerging evidence shows that REM sleep plays a causal role in extinction learning, emotion regulation and consolidation of emotionally positive memories. By using targeted memory reactivation (TMR), a known method where a sound S1 is associated with a waking experience (i.e., a positive outcome of imagery rehearsal therapy in this study) and strengthening it during REM sleep, the investigators want to accelerate the remission of traumatic nightmares and PTSD symptomatology.
  Arms: TMR group
Behavioral: Imagery Rehearsal Therapy — These patients will receive the classic treatment of Imagery Rehearsal Therapy (IRT) for nightmares without association with the sound S1.
  Arms: Control group

SUMMARY:
With this protocol, investigators examine whether targeted memory reactivation (TMR), a technique used to strengthen memories, can accelerate remission of traumatic nightmares and post-traumatic stress disorder (PTSD) symptomatology. This protocol uses TMR during REM sleep to strengthen positive memories generated by Imagery Rehearsal Therapy (IRT), a recommended treatment of nightmares. Patients with PTSD are asked to perform 3 weekly IRT sessions and, while they generate a positive outcome of their recurrent nightmare, half of the patients are exposed to a sound S1 (TMR group), while the other half is not exposed to this sound (control group). All patients will perform IRT every evening at home and will be exposed to the sound S1 during REM sleep with a wireless headband, which automatically detects sleep stages. Clinical evaluation of the severity of PTSD and nightmares before and after (1-month follow-up and 3-months follow-up) this intervention takes place using the validated Clinically Administered PTSD Scale for DSM-5 (CAPS-5, primary outcome measure). The investigators hypothesize that patients treated with IRT and who are exposed, during REM sleep to a sound that had previously been associated with the new positive dream scenario of IRT (TMR group), will have more reduced frequency of PTSD severity and nightmares compared to participants with stimulation of the same, but non-associated, sound during REM sleep (control group).

ELIGIBILITY:
Inclusion Criteria:

* with untreated persistent PTSD according to DSM-5 (> 1 month), suffering from chronic nightmares
* with no active specific treatment for PTSD

Exclusion Criteria:

* patients with active specific treatment for PTSD
* patients with neurological disorders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Clinician-Administered PTSD Scale for DSM-5 | 1 month
  Validated questionnaire that assesses PTSD symptoms, the score ranges from 0-80, zero indicating no symptom severity and 80 indicating the higher symptom severity.
Clinician-Administered PTSD Scale for DSM-5 | 3 months
  Validated questionnaire that assesses PTSD symptoms, the score ranges from 0-80, zero indicating no symptom severity and 80 indicating the higher symptom severity.

SECONDARY OUTCOMES:
Nightmare Frequency | 1 month
  Number of nightmares per week
Nightmare Frequency | 3 months
  Number of nightmares per week
Nightmare Distress Questionnaire | 1 month
  Validated self-report scale to assess the emotional disturbance attributed to the nightmares, the score ranges from 0-52, zero indicating no symptom severity and 52 indicating the higher symptom severity.
Nightmare Distress Questionnaire | 3 months
  Validated self-report scale to assess the emotional disturbance attributed to the nightmares, the score ranges from 0-52, zero indicating no symptom severity and 52 indicating the higher symptom severity.
Positive emotions in dreams | 1 month
  Use of a dream diary
Positive emotions in dreams | 3 months
  Use of a dream diary
PTSD Checklist for DSM5 | 1 month
  Validated self-report measure of PTSD, the score ranges from 0-80, zero indicating no symptom severity and 80 indicating the higher symptom severity.
PTSD Checklist for DSM5 | 3 months
  Validated self-report measure of PTSD, the score ranges from 0-80, zero indicating no symptom severity and 80 indicating the higher symptom severity.
Beck Depression Inventory | 1 month
  Validated self-report scale to assess depressive symptoms, the score ranges from 0-63, zero indicating no symptom severity and 63 indicating the higher symptom severity.
Beck Depression Inventory | 3 months
  Validated self-report scale to assess depressive symptoms, the score ranges from 0-63, zero indicating no symptom severity and 63 indicating the higher symptom severity.
Pittsburgh Sleep Quality Index | 1 month
  Validated self-report scale to assess the quality of sleep, the score ranges from 0-21, zero indicating no symptom severity and 21 indicating the higher symptom severity.
Pittsburgh Sleep Quality Index | 3 months
  Validated self-report scale to assess the quality of sleep, the score ranges from 0-21, zero indicating no symptom severity and 21 indicating the higher symptom severity.

OTHER OUTCOMES:
Sleep efficiency | 1 month
  The ratio between total sleep time and total bed time
REM arousal index | 1 month
  The ratio between number of arousals in stage REM x 60 and REM duration
Arousal index | 1 month
  The ratio between number of arousals in sleep x 60 and sleep duration

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Sleep Medicine, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No